CLINICAL TRIAL: NCT07158372
Title: Research on Identifying Critical Surgical Anatomy in Cholecystectomy Videos Based on Deep Learning
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Capital Medical University (Other); Beijing Anzhen Hospital (Other); Shanghai East Hospital of Tongji University (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Di Dong, Professor, Chinese Academy of Sciences
Other Study IDs: CASMI007
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cholecystectomy; Surgical Video Identification
Keywords: Surgical Video Identification; Deep Learning; Cholecystectomy; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We are collecting laparoscopic cholecystectomy videos and related information. We plan to collect 2,000 retrospective and 200 prospective cases. Enrollment is limited to patients aged 18 years and older diagnosed with laparoscopic cholecystectomy. We will collect information such as laparoscopic cholecystectomy videos and procedure type, excluding patients who did not undergo surgery at the original hospital or whose videos were blurry.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- The First Affiliated Hospital of Zhengzhou University: patients aged 18 years and older diagnosed with laparoscopic cholecystectomy. We will collect information such as laparoscopic cholecystectomy videos and procedure type, excluding patients who did not undergo surgery at the original hospital or whose videos were blurry.
  Interventions: Diagnostic Test: AI-assisted Intraoperative Anatomy Analysis
- Beijing Luhe Hospital, Capital Medical University: patients aged 18 years and older diagnosed with laparoscopic cholecystectomy. We will collect information such as laparoscopic cholecystectomy videos and procedure type, excluding patients who did not undergo surgery at the original hospital or whose videos were blurry.
  Interventions: Diagnostic Test: AI-assisted Intraoperative Anatomy Analysis
- Shanghai East Hospital of Tongji University: patients aged 18 years and older diagnosed with laparoscopic cholecystectomy. We will collect information such as laparoscopic cholecystectomy videos and procedure type, excluding patients who did not undergo surgery at the original hospital or whose videos were blurry.
  Interventions: Diagnostic Test: AI-assisted Intraoperative Anatomy Analysis
- Peking university people's hospital: patients aged 18 years and older diagnosed with laparoscopic cholecystectomy. We will collect information such as laparoscopic cholecystectomy videos and procedure type, excluding patients who did not undergo surgery at the original hospital or whose videos were blurry
  Interventions: Diagnostic Test: AI-assisted Intraoperative Anatomy Analysis

INTERVENTIONS:
Diagnostic Test: AI-assisted Intraoperative Anatomy Analysis — This is a prospective study on patients aged 18 years or more diagnosed with laparoscopic cholecystectomy. We will collect information such as laparoscopic cholecystectomy videos and procedure type, excluding patients who did not undergo surgery at the original hospital or whose videos were blurry.

SUMMARY:
Laparoscopic cholecystectomy is a common surgical procedure, but it carries the potential for bile duct injury and other surgical risks. To provide visual assistance to surgeons during surgery and mitigate these risks, this research project aims to develop a real-time object recognition algorithm based on deep learning technology. This algorithm will label key anatomical structures in laparoscopic cholecystectomy videos, providing surgeons with immediate information on dangerous and safe areas.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is a common surgical procedure, but it carries the potential for bile duct injury and other surgical risks. To provide visual assistance to surgeons during surgery and mitigate these risks, this research project aims to develop a real-time object recognition algorithm based on deep learning technology. This algorithm will label key anatomical structures in laparoscopic cholecystectomy videos, providing surgeons with immediate information on dangerous and safe areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or above who are diagnosed by a doctor as needing laparoscopic cholecystectomy

Exclusion Criteria:

* Patients who did not undergo surgery at the original hospital and those whose videos were blurry were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or above who are diagnosed by a doctor as needing laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Dice Similarity Coefficient | 3 years
  Dice Similarity Coefficient is a statistical measure of the similarity between two sets of data. In the context of image segmentation, it is used to quantify the spatial overlap between a predicted segmentation mask and its corresponding ground truth mask.
Mean Intersection over Union | 3 years
  Mean Intersection over Union provides a measure of the overlap between the predicted segmentation and the ground truth, averaged across all classes present in the dataset.
Global Accuracy | 3 years
  The proportion of correctly classified pixels out of the total number of pixels in the image.

SECONDARY OUTCOMES:
Inference Latency | 3 years
  time taken by the algorithm to process a single video frame and generate the segmentation masks (inference latency), or equivalently, the number of frames processed per second

OTHER OUTCOMES:
Class-Specific Precision and Recall for Critical Structures | 3 years
  Precision: The proportion of predicted pixels for a structure that are actually part of that structure Recall: The proportion of actual ground truth pixels for a structure that were correctly identified by the algorithm

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - Peking university people's hospital, Beijing
  - Shanghai East Hospital of Tongji University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided